CLINICAL TRIAL: NCT01877200
Title: A Cross-Sectional Survey to Evaluate Diabetes Management, Control, Complications, Psychosocial Aspects of Patients With Type 2 Diabetes in Bangladesh
Acronym: DiabCare Asia
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-4071; U1111-1137-2729 (Other: WHO)
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with diabetes (type 2)
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Patients will fill out a questionnaire by interview.

SUMMARY:
This study is conducted in Asia. The aim of this non-interventional study is to evaluate the the current status of diabetes management, control, and complications in diabetic subjects with type 2 diabetes in Bangladesh.

ELIGIBILITY:
Inclusion Criteria:

* People with type 2 diabetes mellitus (DM) who are being treated, with any of the non-pharmacological or pharmacological options, at a particular centre for at least 1 year and who have visited the centre within the last 3-6 months
* Patients willing to sign informed consent form

Exclusion Criteria:

* Previous participation in this study
* Unable to comply with protocol requirements
* Confirmed or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People treated for at least a year are eligible for the study. The selection of the patients will be done randomly by the individual physician involved in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2092 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients having HbA1c ((Glycosylated Haemoglobin) as measured during survey) less than 7% | Evaluated at the first visit (only one study visit)

SECONDARY OUTCOMES:
Mean Fasting Plasma Glucose (FPG) of patients | Evaluated at the first visit (only one study visit)
Mean Postprandial Plasma Glucose (PPG) of patients | Evaluated at the first visit (only one study visit)
Mean HbA1c of patients | Evaluated at the first visit (only one study visit)
Proportion of patients having dyslipidemia and hypertension | Evaluated at the first visit (only one study visit)
Proportion of patients having cardiovascular complications | Evaluated at the first visit (only one study visit)
Proportion of patients having peripheral vascular disease | Evaluated at the first visit (only one study visit)
Proportion of patients having diabetic nephropathy | Evaluated at the first visit (only one study visit)
Proportion of patients having diabetic eye complications | Evaluated at the first visit (only one study visit)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Dhaka, Bangladesh

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com